CLINICAL TRIAL: NCT01949402
Title: Thoracic Ultrasonography in the Assessment of Extravascular Lung Water & Respiratory Failure
Brief Title: A New Way of Looking at Your Lungs
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: TUS-EVLW1
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Respiratory Failure; Acute Dyspnoea
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Haemodialysis: Patients with end-stage renal failure (ESRF) requiring long-term regular haemodialysis.
  Interventions: Other: Computed Tomography; Other: Thoracic ultrasound; Other: Spirometry; Other: Blood tests
- Chronic Obstructive Pulmonary Disease: Patients with a confirmed diagnosis of COPD based on clinical history, obstructive spirometry (FEV1/VC ratio <70%) and radiology (e.g. hyperexpansion on plain chest radiograph; evidence of small airways disease or emphysema on cross-sectional imaging).
  Interventions: Other: Computed Tomography; Other: Thoracic ultrasound; Other: Spirometry; Other: Blood tests
- Interstitial Lung Disease: Patients with a confirmed diagnosis of ILD based on clinical history and radiology (evidence of ILD on cross-sectional imaging).
  Interventions: Other: Computed Tomography; Other: Thoracic ultrasound; Other: Spirometry; Other: Blood tests
- Control: Age-matched healthy volunteers with no history of cardiac, respiratory or renal disease.
  Interventions: Other: Computed Tomography; Other: Thoracic ultrasound; Other: Spirometry; Other: Blood tests

INTERVENTIONS:
Other: Computed Tomography — The CT scan will be performed on a 16 slice GE Discovery 670 SPECT CT scanner. A slice thickness of 0.625mm will be used. Images are acquired during an inspiratory breath hold of up to 20 seconds to minimise movement artefact. The patient will be lying supine and the scan will be a non-contrast study. Using a low dose CT chest protocol (1.7 mSv) will minimise the exposure to ionising radiation of study participants.
  Participants in the haemodialysis arm of the study will have a CT done before and after haemodialysis. Participants in all other arms will have a single CT scan done during their study "visit".
Other: Thoracic ultrasound — The ultrasound will be performed by a single operator. The patient's position will ideally be with the patient sitting up at 45°. Ultrasound images and clips will be recorded at 10 points over each hemithorax - the 2nd, 4th and 6th intercostal spaces (ICS) in the mid-clavicular line; the 2nd, 4th and 6th ICS in the mid-axillary line; and the 2nd, 5th, 7th and 9th ICS posteriorly. Ultrasound estimation of the height of the right internal jugular vein will be undertaken. Central venous pressure will be calculated by adding 5cm. Inferior vena cava diameter will also be measured at end-inspiration and expiration. The time taken to perform each ultrasound will be recorded. Control, COPD and ILD groups will be scanned on a single occasion. Haemodialysis group will have 4 scans.
Other: Spirometry — All participants in the study will undergo basic spirometry as specified in the study assessments. This is considered a low-risk intervention and no harm is expected as a consequence of participation in the study.
Other: Blood tests — All participants in the study will undergo blood tests as specified in the study assessments. This is considered a low-risk intervention and no harm is expected as a consequence of participation in the study.

SUMMARY:
There is increasing interest in how thoracic (chest) ultrasound might enhance the management of patients with respiratory failure and breathlessness, particularly in the emergency admissions or intensive care setting. Thoracic ultrasound is already used in a number of clinical settings. It is recognised that a number of lung abnormalities can be identified using thoracic ultrasound, such as consolidation (in pneumonia) or peripheral soft tissue lesions (in lung cancer). Furthermore, thoracic ultrasound offers clinicians a non-invasive diagnostic tool that provides immediate feedback and results.

Patients with breathlessness and respiratory failure represent a significant proportion of emergency admissions to hospital and commonly require urgent treatment with limited information available to guide the clinician. The range of diseases that present with breathing difficulties is broad (e.g. pneumonia, heart failure, pulmonary embolus) and difficult to differentiate in patients who often have multiple medical problems. This leads to non-specific treatment in the face of diagnostic uncertainty with the associated risks of treatment complications, increased morbidity and mortality, and distress for patients and relatives. It is in the assessment of these patients with acute respiratory failure where thoracic ultrasound might be of greatest benefit and which this research is designed to address.

This is a single centre study (Churchill Hospital, Oxford) recruiting 125 participants over an eight month period. The study will test the reliability of a thoracic ultrasound protocol at identifying lung abnormalities in a stable outpatient population with respiratory disease (chronic obstructive pulmonary disease; interstitial lung disease; patients on haemodialysis to replicate acute pulmonary oedema / heart failure). It is hoped the results of this study will inform further research in acutely unwell patients with respiratory failure and breathlessness to see whether thoracic ultrasound can improve diagnostic and therapeutic decisions.

DETAILED DESCRIPTION:
This is a prospective cohort study and forms part of educational research intended to ultimately contribute towards a higher degree (MD or DPhil). The study is being co-ordinated through the Oxford Respiratory Trials Unit, Churchill Hospital, Oxford and has been developed by the study co-ordinator (Dr Corcoran) and Chief Investigator (Dr Rahman) with support from Professor Gleeson.

This study will assess the efficacy of TUS in identifying extravascular lung water (EVLW) through the presence or absence of B-lines (also known as "comet tails") on ultrasound; whilst also determining whether TUS can distinguish between other pulmonary pathologies that may cause both a similar ultrasonographic appearance and respiratory compromise. A TUS protocol will be tested and validated in a stable patient population, concurrently assessing patient and operator satisfaction with the tool. It is intended that the results of this study will inform a larger second-phase study of a modified TUS protocol in the acute clinical setting (medical admissions unit +/- emergency department).

Potential participants in this study will be screened from normal clinical care in the relevant departments at the Churchill Hospital, Oxford - i.e. specialist COPD and ILD clinics in the respiratory department; outpatient haemodialysis units in the renal department. Healthy volunteers will also be sought using advertisements placed on noticeboards in the Oxford University Hospitals NHS Trust and selected Oxford University departments.

All participants enrolled in the study will undergo CT and thoracic ultrasound scanning as per the study protocol. These are low-risk interventions with no harm expected as a direct consequence of participation in the study.

Participants will also undergo baseline spirometry (if not done in the last month) and blood tests for the purposes of the study; these are also considered low-risk interventions with no harm expected as a direct consequence of participation in the study.

The study involves only a single visit and therefore it should impose a minimal burden on participants, and for the majority of participants their study visit will be arranged to coincide with a pre-arranged trip to the hospital for normal clinical care (e.g. a regular haemodialysis or outpatient clinic visit).

ELIGIBILITY:
Inclusion Criteria:

* Haemodialysis (n=50) - patients with end-stage renal failure (ESRF) requiring long-term regular haemodialysis.
* Chronic Obstructive Pulmonary Disease (COPD) (n=25) - patients with a confirmed diagnosis of COPD based on clinical history, obstructive spirometry (FEV1/VC ratio <70%) and radiology (e.g. hyperexpansion on plain chest radiograph; evidence of small airways disease or emphysema on cross-sectional imaging).
* Interstitial Lung Disease (ILD) (n=25) - patients with a confirmed diagnosis of ILD based on clinical history and radiology (evidence of ILD on cross-sectional imaging).
* Control (n=25) - age-matched healthy volunteers with no history of cardiac, respiratory or renal disease.

Exclusion Criteria:

* Age < 18 years
* Inability to provide informed consent to participate in the study
* Pregnant or breastfeeding
* Known diagnosis of heart failure or chronic renal failure in participants recruited to the COPD or ILD arms of the study.
* Known diagnosis of COPD or ILD in participants recruited to the haemodialysis arm of the study.
* Known history of cardiac, respiratory or renal disease in participants recruited to the control arm of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be screened from normal clinical care in the outpatient haemodialysis unit and specialist respiratory clinics (COPD and ILD) at the Churchill Hospital, Oxford. Age-matched volunteers will also be sought for the control arm of the study.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2014-02; Primary Completion 2016-07-31 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
The total lung ultrasound B-line score. | At enrollment (1 single visit only)
  The total lung ultrasound B-line score (representing the presence of extravascular lung water) and changes in overall fluid status during haemodialysis.

SECONDARY OUTCOMES:
Lung ultrasound identification of B-lines and differentiation between extravascular lung water | At enrollment (1 single visit only)
  Lung ultrasound identification of B-lines and differentiation between extravascular lung water (EVLW) and other causes of this ultrasonographic appearance.
The lung ultrasound B-line score at differing anatomical locations around the thoracic cage | at enrollment (1 single visit only)
  The lung ultrasound B-line score (representing the presence of EVLW) at differing anatomical locations around the thoracic cage and changes in overall fluid status during haemodialysis.
The total lung ultrasound B-line score | At enrollment (1 single visit only)
  The total lung ultrasound B-line score (representing the presence of EVLW) and changes in patient breathlessness as measured by a visual analogue scale during haemodialysis.
Patient satisfaction with the thoracic ultrasound protocol | At enrollment (1 single visit only)
  Patient satisfaction with the thoracic ultrasound protocol as measured using a Likert-type scale.

CONTACTS AND LOCATIONS:
Overall Officials: Najib Rahman, DPhil, Study Chair — University of Oxford; John Corcoran, BM BCh, Principal Investigator — University of Oxford; Fergus Gleeson, Prof, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- Oxford Respiratory Trials Unit, Oxford, United Kingdom